CLINICAL TRIAL: NCT04322773
Title: Effectiveness of Interleukin-6 Receptor Inhibitors in the Management of Patients With Severe SARS-CoV-2 Pneumonia: An Open-Label, Multicenter Sequential and Cluster Randomized Trial
Brief Title: Anti-il6 Treatment of Serious COVID-19 Disease With Threatening Respiratory Failure
Acronym: TOCIVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated due to changed clinical conditions and too few patients available
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APPI2-CV-2020-01
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Corona Virus Disease
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Roactemra iv (Experimental): Single dose treatment with 400 mg tocilizumab intravensously
  Interventions: Drug: RoActemra iv; Other: Standard medical care
- Roactemra sc (Experimental): Single dose treatment with 2 x 162 mg tocilizumab subcutaneously
  Interventions: Drug: RoActemra sc; Other: Standard medical care
- Kevzara sc (Experimental): Single dose treatment with 1 x 200 mg sarilumab subcutaneously
  Interventions: Drug: Kevzara sc; Other: Standard medical care
- Standard care (Active Comparator): Management as usual
  Interventions: Other: Standard medical care

INTERVENTIONS:
Drug: RoActemra iv — single dose treatment with tocilizumab 400 mg intravenously
  Other Names: tocilizumab 400 mg
  Arms: Roactemra iv
Drug: RoActemra sc — single dose treatment with tocilizumab 2 x 162 mg subcutaneously
  Other Names: tocilizumab 2 x 162 mg
  Arms: Roactemra sc
Drug: Kevzara sc — single dose treatment with sarilumab 1 x 200 mg subcutaneously
  Other Names: sarilumab 1 x 200 mg
  Arms: Kevzara sc
Other: Standard medical care — management as usual

SUMMARY:
Coronavirus disease 2019 (COVID-19) is caused by the newly discovered coronavirus, SARS-CoV-2. The median time from onset of symptoms of COVID-19 to development of acute respiratory distress syndrome (ARDS) has been reported as short as 9 days. No effective prophylactic or post-exposure therapy is currently available. According to data from the Danish Health Authority (www.sst.dk/corona), as of March 21st, 2020, there were 1326 patients infected with the disease in Denmark, more than 250 are admitted to a hospital, and >50 of them have required intensive care. Nearly 350.000 cases and 15.000 deaths have been reported globally. These numbers are likely to markedly increase during the coming weeks, challenging the capacity of health systems worldwide.

In patients infected with SARS-CoV-2, it has been described that disease severity and outcomes are related to the characteristics of the immune response. Interleukin (IL)-6 and other components of the inflammatory cascade contribute to host defense against infections. However, exaggerated synthesis of IL-6 can lead to an acute severe systemic inflammatory response known as 'cytokine storm'. In the pathogenesis of SARS-CoV-2 pneumonia, a study found that a cytokine storm involving a considerable release of proinflammatory cytokines occurred, including IL-6, IL-12, and tumor necrosis factor α (TNF-α). Studies on the Middle East respiratory syndrome caused by another coronavirus (MERS-CoV), indicate that cytokine genes of IL-6, IL-1β, and IL-8 can be markedly upregulated. Similarly, patients with SARS-CoV-2 pneumonia admitted to an intensive care unit had higher plasma levels of cytokines including IL-6, IL-2, IL-7, IL-10, granulocyte-colony stimulating factor (G-CSF), interferon-γ-inducible protein (IP10), monocyte chemoattractant protein (MCP1), macrophage inflammatory protein 1 alpha (MIP1A), and TNF-α. These findings indicate that the magnitude and characteristics of the cytokine response is related to the severity and prognosis of patients with SARS-CoV-2 pneumonia.

It has been suggested that IL-6 blockade may constitute a novel therapeutic strategy for other types of cytokine storm, such as the systemic inflammatory response syndrome including sepsis, macrophage activation syndrome and hemophagocytic lymphohistiocytosis. Remarkable beneficial effects of IL-6 blockade therapy using a IL-6 receptor inhibitor has been described in patients with severe SARS-CoV-2 pneumonia in a retrospective case series from China.

Currently, there are two available drugs based on human monoclonal antibodies against IL-6 receptor, tocilizumab (RoActemra, Roche) and sarilumab (Kevzara, Sanofi). IL-6 receptor inhibitors are currently licensed for several autoimmune disorders and are considered well tolerated and safe in general. The most common side effects reported are upper respiratory tract infections, headache, hypertension, and abnormal liver function tests. The most serious side effects are serious infections, complications of diverticulitis, and hypersensitivity reactions.

it is hypothesized that IL-6 might play a key role in the cytokine storm associated with serious adverse outcomes in patients infected with SARS-CoV-2 pneumonia, and that blockade of IL-6 would be suitable therapeutic target for these patients. The study will investigate the effect of different types of IL-6 inhibition versus no adjuvant treatment compared to standard of care in patients with severe SARS-CoV-2 pneumonia.

Primary objective: To compare the effect of either one of three IL-6 inhibitor administrations, relative to the standard of care, on time to independence from supplementary oxygen therapy, measured in days from baseline to day 28, in patients with severe SARS-CoV-2 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed by real time-PCR and
* Positive imaging: consolidation, ground glass opacities, or bilateral pulmonary infiltration either by CT-scan or chest x-ray; and
* Need of oxygen therapy to maintain SO2>94% OR FiO2/PaO2 > 20 and at least two of the following laboratory measures:
* CRP level >70 mg/L
* CRP level >= 40 mg/L and doubled within 48 hours (without other confirmed infectious or non-infectious course),
* Lactatdehydrogenase > 250 U/L,
* thrombocytopenia < 120.000 x 10E9/L,
* lymphocyte count < 0.6 x 10E9/L,
* D-dimer > 1 ug/mL,
* serum ferritin > 300 ug/mL

Exclusion Criteria:

* pregnancy suspected or confirmed,
* severe heart failure,
* suspected or confirmed bacterial infection,
* current solid or hematological malignancy,
* neutropenia,
* ALAT elevation more than three times the laboratory upper limit,
* ASA class 5 (after COVID19 admission) or higher at inclusion (prior admission),
* severe chronic obstructive pulmonary disease or heart failure (NYHA class II or higher),
* pregnant or lactating women,
* current treatment with conventional synthetic disease-modifying antirheumatic drugs (DMARDs)/immunosuppressive agents including IL-6 inhibitors, or with Janus kinase inhibitors (JAKi) in the past 30 days or plans to receive during the study period,
* current use of chronic oral corticosteroids in a dose higher than prednisone 10 mg or equivalent per day,
* previous or active tuberculosis (TB),
* HIV infection regardless of immunological status, hepatitis,
* evidence of recent (30 days) invasive bacterial or fungal infections,
* patients who have received immunosuppressive antibody therapy within the past 5 months, including intravenous immunoglobulin or plans to receive during the study period,
* IV drug abuse,
* history of inflammatory bowel disease,
* diverticulitis,
* ulcer,
* perforated gastrointestinal tract,
* participation in any clinical research study evaluating an investigational product (IP) or therapy within 3 months and less than five half-lives of IP prior inclusion to the study,
* any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study,
* inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Time to independence from supplementary oxygen therapy | days from enrolment up 28 days

SECONDARY OUTCOMES:
Number of deaths | 28 days from enrolment
Days out of hospital and alive | 28 days from enrolment
Ventilator free days alive and out of hospital | 28 days from enrolment
C-reactive protein (CRP) level | baseline
  Measured from standard blood test
C-reactive protein (CRP) level | peak during hospitalisation, up to 28 days
  Measured from standard blood test
C-reactive protein (CRP) level | 14 days
  Measured from standard blood test
C-reactive protein (CRP) level | 28 days
  Measured from standard blood test
Number of participants with serious adverse events | During treatment, up to 28 days
  Measured as occurrence of any serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lars Erik Kristensen, PhD, Principal Investigator — The Parker Institute
Locations (2):
- Denmark (2):
  - Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Hillerød Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code